CLINICAL TRIAL: NCT02161705
Title: Pre-operative Paravertebral Blocks to Decrease Post-operative Pain Following Mastectomy With Immediate Tissue Expander Reconstruction
Brief Title: Pre-op Paravertebral Blocks to Decrease Post-op Pain Following Mastectomy With Immediate Tissue Expander (TE) Reconstruction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual due to change in standard of care procedure.
Sponsor: Johns Hopkins University (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00075957; 311945 (Other Grant/Funding Number: Plastic Surgery Education Foundation)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Quality of Life
Keywords: Immediate breast reconstruction; pain control; post mastectomy pain control
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Agnosia | interventions — Ropivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine Group (Experimental): Paravertebral block injections of study solution will occur using the landmark-based classic technique with a 22-gauge Tuohy needle to deliver 0.5% ropivacaine (up to 0.8 mL/kg, equivalent to 4mg/kg).
  Interventions: Drug: Ropivacaine
- Saline Group (Placebo Comparator): Paravertebral block injections of normal saline (up to 0.8 mL/kg) will occur using the landmark-based classic technique with a 22-gauge Tuohy needle. Immediately after completion of the injections, patients will be repositioned supine and general anesthesia induced in the standard manner.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — 0.5% ropivacaine (up to 0.8 mL/kg, equivalent to 4mg/kg) administered in paravertebral block
  Other Names: Naropin
  Arms: Ropivacaine Group
Drug: Saline — Up to 0.8 mL/kg of normal saline administered
  Other Names: Normal Saline
  Arms: Saline Group

SUMMARY:
Primary Objective To determine if post-operative static pain scores differ between women undergoing bilateral mastectomy followed by bilateral immediate tissue expander reconstruction randomized either to ropivacaine- (treatment) or saline- (placebo) pre-operatively placed paravertebral blocks.

Post-operative pain scores will be measured by a 0-10 Likert scale 6 hours after the end of surgery while the patient is still hospitalized (post-operative day 0). This will be patient-provided data. Unblinded data analysis will compare scores between treatment and control groups.

Secondary Objectives To determine if post-operative moving pain scores, opioids use, nausea, and sleep interference differ between women undergoing bilateral mastectomy followed by bilateral immediate tissue expander reconstruction randomized either to ropivacaine- (treatment) or saline- (placebo) pre-operatively placed paravertebral blocks.

Pain score, opioids use, nausea, and sleep interference data will be collected via patient self-report. When possible (i.e., while hospitalized) objective data on opioids and other pain medication administered to the patient will be used.

Tertiary Objectives To determine if long-term changes in Quality of Life scores [the RAND-36 Health Survey, Disability of the Arm, Shoulder, and Hand (Quick DASH) questionnaire, and Breast-Q scores] differ between women undergoing bilateral mastectomy followed by bilateral immediate tissue expander reconstruction randomized either to ropivacaine- (treatment) or saline- (placebo) pre-operatively placed paravertebral blocks.

This data will be collected via validated questionnaires through patient interviews at 3-months, 2-years, and 4-years (±14 days) after surgery.

Once enrolled in the study, participants will be encouraged to remain in the study for the 4 years following surgery in order to get final pain scores and quality-of-life/health outcome survey information. Participants who cannot be contacted after several phone attempts and the sending of 2 certified letters via US Postal Service for 3-month, 2-year, and/or 4-year outcome assessments will be considered lost to follow-up.

DETAILED DESCRIPTION:
This double-blind, randomized, controlled clinical trial comparing patient-reported pain and pain medication/narcotic use between patients randomized to treatment (ropivacaine) or placebo (saline) delivered via paravertebral block to the mastectomy site. Candidates will have chosen to have a mastectomy on one side immediately followed with tissue expander placement breast reconstruction.

Patients will be randomized 1:1 to ropivacaine- (treatment) or saline-(placebo) paravertebral blocks in a double-blinded design. Patient-specific surgical details will be recorded intraoperatively. Following the surgery, post-operative pain, pain medication/opioid use, and the occurrence of adverse events (AEs)/serious adverse events (SAEs) will be assessed on Days 1, 2, and 3. A clinic visit occurs on Day 7 when additional data are collected (updated medical history, pain medication/opioid use, AEs/SAEs, and study questionnaires. Using two pain scales, the Patient Pain Assessment Questionnaire (Appendix A) and Subjective Pain Survey (Appendix B), the post-operative pain will be compared between treatment and control groups. Differences in opioids use between groups at different time points will also be assessed as a more objective measure of post-operative pain.

Long-term quality-of-life/health outcomes assessments will be done on post-operative Day 90 (±14 days), Year 2 (±14 days), and Year 4 (±14 days). The Year 2 and Year 4 follow-ups are included as tertiary endpoints to capture differences in chronic pain, and patients will be asked to complete the same questionnaires as at the Day 90 follow up.

The investigators hypothesize that post-operative static pain scores will be lower in ropivacaine patients vs. placebo patients in women undergoing mastectomy and immediate reconstruction with placement of tissue expanders. We believe that post-operative moving pain scores, opioids use, nausea, and sleep interference will be likewise improved. We further hypothesize that this decreased post-operative pain may lead to improvements in long-term health outcomes as measured by validated questionnaires. In the presence of clear need and lack of published studies regarding this precise patient population, it is important to determine if paravertebral blocks do reduce post-operative pain, and improve opioids use, nausea, sleep interference, and length of hospital stay in patients undergoing immediate tissue expander breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Be Female aged 18-100 years.
* Choose mastectomy followed by bilateral immediate tissue expander breast reconstruction.
* Have no inflammatory breast cancers.
* Be aware of the nature of her malignancy.
* Understand the study purpose, requirements, and risks.
* Be able and willing to give informed consent.

Exclusion Criteria:

* Any concurrent opioid analgesic use (baseline opioid use must be 0 to be eligible).
* Liver dysfunction and/ or cirrhosis.
* Renal insufficiency, with creatinine greater than 1.5 mg/mL.
* Patients weighing less than 50 Kg.
* Concurrent use of the SSRI antidepressant fluvoxamine (Luvox).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gedge D Rosson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Group | Saline Group
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Group | Saline Group | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 50 [42.5 to 59] | 54 [47 to 57] | 53.5 [43.75 to 57.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Subjective Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — The Subjective Pain Assessment tool is a likert scale model tool (e.g. 0-5, 0-10) which asks patients to score their perception of how painful a particular act is (e.g How painful is biting your tongue?) on a scale of 0-5, from a preset list of questions regarding pain. This is used to establish a baseline value for a patients pain threshold. Population: 3 patients in the Saline group did not fill out subjective pain score assessments.
  units on a scale
    number analyzed (Participants) | 9 | 6 | 15
    (all) | 3.38 [2.69 to 3.50] | 3.69 [2.75 to 4.16] | 3.38 [2.75 to 3.88]
Static Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — Static pain score assesses a patient's perception of pain when they are not moving. Patients rate this pain on a scale of 0-10, where 0 represents no pain and 10 represents the worst pain the patient has experienced.
  units on a scale | 0 [0 to 1] | 0 [0 to 4.5] | 0 [0 to 1]
Moving Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — Moving pain score assesses a patient's perception of pain when they are moving. Patients rate this pain on a scale of 0-10, where 0 represents no pain and 10 represents the worst pain the patient has experienced.
  units on a scale | 0 [0 to 6] | 0 [0 to 9] | 0 [0 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Static Pain Score
Description: To determine if post-operative static pain scores differ between women undergoing bilateral mastectomy followed by bilateral immediate tissue expander breast reconstruction randomized either to ropivacaine- (treatment) or saline- (placebo) pre-operatively placed paravertebral blocks.
  Post-operative pain, pain medication/narcotic use, and assessment for adverse events (AEs)/serious adverse events (SAEs) will be assessed the Day of surgery through post-operative Day 7. A clinic visit occurs on Day 7 where additional data collected (updated medical history, pain medication/narcotic use, AEs/SAEs, and study questionnaires).
  Static pain refers to pain when the patient is at rest. Patients report pain on a scale of 0-10 were in 0 represents no pain and 10 the most severe pain they have experienced.
Time Frame: Day of Surgery through Day 7
Population: 1 Patient in the saline group was lost to follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine Group | Saline Group
Number analyzed (Participants) | 9 | 8
units on a scale | 1.5 [0.63 to 3.19] | 1 [0.09 to 2.5]

2. Secondary Outcome: Quality of Life Scores as Assessed by the BREAST-Q Score
Description: To determine if long-term changes in Quality of Life scores [BREAST-Q scores] differ between women undergoing mastectomy followed by immediate tissue expander reconstruction randomized either to ropivacaine- (treatment) or saline- (placebo) pre-operatively placed paravertebral blocks.
  The BREAST-Q score questionnaire items in each scale are arranged in a clinically relevant hierarchy (e.g., Satisfaction with Breasts scale ranges from "How satisfied are you with how you look in a mirror clothed?" to "How satisfied are you with how you look in the mirror unclothed?"). Scores will range from 0-100. Lower scores indicate lower quality of life and vice versa.
  This data will be collected via validated questionnaires through patient interviews at 1-month, 3-months, 2-years, and 4-years (±14 days) after surgery.
  Once enrolled in the study, participants will be encouraged to remain in the study for the 4 years following surgery in order to get final pain scores and quality-of-life/heal
Time Frame: Postoperative Day-30, Day-90 , 2-years, and 4-years (±14 days) after surgery.
Population: The minimum data needed to assess this outcome measure was not collected for any participant and thus could not be analyzed for any of the participants.
Arm/Group | Ropivacaine Group | Saline Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Description: No of the procedures are experimental or new. The novelty of the study simply is the use of the paravertebral block in patients undergoing breast reconstruction.
Arm/Group | Ropivacaine Group | Saline Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02161705/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02161705/Prot_SAP_001.pdf